CLINICAL TRIAL: NCT00604890
Title: Dose-Ranging Clinical Trial of Topical Creams Containing API 31510 for the Treatment of Superficial Basal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTL0108
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2019-02

CONDITIONS: Superficial Basal Cell Carcinoma
Keywords: Double-Blind; Placebo; Topical; Treatment; Dose-Ranging; sBCC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 (Experimental): Active cream, 3% AM & PM
  Interventions: Drug: API 31510 3% Topical Cream
- 2 (Placebo Comparator): Placebo cream AM ; 3% active cream PM
  Interventions: Drug: API 31510 3% Topical Cream; Other: Placebo
- 3 (Placebo Comparator): Placebo cream AM; 1.5% active cream PM
  Interventions: Drug: API 31510 1.5% Topical Cream; Other: Placebo
- 4 (Placebo Comparator): Placebo AM and PM
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: API 31510 3% Topical Cream — Topical treatment 3% active cream applied to the lesion
  Arms: 1; 2
Drug: API 31510 1.5% Topical Cream — Topical treatment 1.5% active cream applied to the lesion
  Arms: 3
Other: Placebo — Topical treatment placebo applied to the lesion
  Arms: 2; 3; 4

SUMMARY:
The purpose of this study is to determine the safety and tolerability of pharmaceutical compound (API 31510) topical cream topically applied to superficial basal cell carcinomas to obtain preliminary efficacy data for the treatment of superficial basal cell carcinomas by API 31510 topical cream. The study population will include one hundred and sixty (160) otherwise healthy male or female adults with one or more histologically confirmed superficial basal cell carcinoma lesions. One target lesion with an area of less than one inch will be designated for study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 18 years of age
* Primary, histologically confirmed sBCC with a minimum area of 0.5 cm2 and with a maximum diameter of 2.0 cm target sBCC lesion suitable for excision
* Histological diagnosis made no more than 4 weeks prior to the screening visit
* Histological biopsy removed 25% or less of the target lesion
* No other dermatological disease in the sBCC target site or surrounding area
* Willing to refrain from using non-approved lotions or creams on the target site and surrounding area during the treatment period. Willing to refrain from washing the treated area for at least 8 hours following the application of study medication
* Willing to refrain from exposure to direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study
* Laboratory values for the tests listed in the Study Schedule on page 2 within the reference ranges as defined by the central laboratory, or "out of range" test results that are clinically acceptable to the investigator.
* Ability to follow study instructions and likely to complete all study requirements
* Written informed consent obtained, including consent for tissue to be examined and stored by the central dermatopathologist
* Written consent to allow photographs of the target sBCC lesion to be used as part of the study data
* For females of childbearing potential, a negative pregnancy test at screening and using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy)

Exclusion Criteria:

* Pregnant or lactating
* Presence of known or suspected systemic cancer
* Histological evidence of nBCC, SCC, or any other tumor in the biopsy specimen
* Histological evidence of severe squamous metaplasia, infiltrative, desomoplastic or micronodular growth patterns in the biopsy specimen
* History of recurrence of the target sBCC lesion
* Evidence of dermatological disease or confounding skin condition in the treatment area, e.g., SCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema, xeroderma pigmentosa
* Concurrent disease or treatment that suppresses the immune system
* Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the patient at undue risk
* Known sensitivity to any of the ingredients in the study medication
* Use of a tanning parlor or other excessive or prolonged exposure to ultraviolet light or direct sunlight during the course of the study
* Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit
* Use of systemic retinoids within the 6 months prior to the screening period
* Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the screening period
* Use of topical immunomodulators within 2 cm of the target BCC lesion within the 4 weeks prior to the screening period
* Treatment with the following topical agents within the 4 weeks prior to the screening visit: levulanic acid, 5-fluorouracil, coricosteroids, retinoids, diclofenac, hyaluronic acid, imiquimod
* Undergone a facial resurfacing procedure, i.e., chemical peel, laser resurfacing, dermabrasion, within the 6 months prior to the screening visit, if the target sBCC lesion is on the face
* Treatment with liquid nitrogen, surgical excision or curettage within 2 cm of the target sBCC lesion during the 4 weeks prior to the screening visit
* Elective surgery within 4 weeks prior to the screening visit, during the study, or 4 weeks after the treatment period
* Evidence of current chronic alcohol or drug abuse
* Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the screening visit
* In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions of the protocol and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wilson, MD, Principal Investigator — Education and Research Foundation
Locations (11):
- United States (11):
  - Burke Pharmaceuticals, Hot Springs, Arkansas
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Colorado Medical Research Center, Denver, Colorado
  - Dermatology Associates and Research, Coral Gables, Florida
  - Gwinnett Clinical Research, Snellville, Georgia
  - Scott D. Glazer, M.D., S.C., Buffalo Grove, Illinois
  - Christie Clinic, Champaign, Illinois
  - Long Island Skin Cancer and Dermatologic Surgery, PC, Smithtown, New York
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Education & Research Foundation, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- 3% Active Cream BID(Twice Daily): Topical Treatment 3.0% active cream applied to the lesion twice daily (BID)
- 3% Active Cream QD(Once Daily): Topical treatment 3.0% active cream applied to the lesion once daily (PM) plus placebo cream applied to the lesion once daily (AM)
- 1.5% Active Cream QD(Once Daily): Topical treatment 1.5% active cream applied to the lesion once daily (PM) plus placebo cream applied to the lesion once daily (AM)
- Placebo BID(Twice Daily): Placebo cream applied to the lesion twice daily
Period: Overall Study
Arm/Group | 3% Active Cream BID(Twice Daily) | 3% Active Cream QD(Once Daily) | 1.5% Active Cream QD(Once Daily) | Placebo BID(Twice Daily)
Started | 47 | 45 | 48 | 46
Completed | 44 | 45 | 47 | 42
Not Completed | 3 | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- 3% BID: 3.0% active twice daily (BID)
- 3% QD: 3.0% active cream once daily (QD) plus placebo cream QD
- 1.5% QD: 1.5% active cream once daily (QD) plus placebo cream QD
- Placebo: Placebo cream twice daily (BID)
- Total: Total of all reporting groups
Arm/Group | 3% BID | 3% QD | 1.5% QD | Placebo | Total
Number analyzed (Participants) | 47 | 45 | 48 | 46 | 186
Age, Continuous [Mean (Full Range); unit: years] | 62.6 [36 to 83] | 61.2 [34 to 84] | 60.4 [34 to 81] | 62.8 [37 to 90] | 61.7 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 23 | 16 | 76
  Male | 30 | 25 | 25 | 30 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: To determine the number of participants with a complete response, defined as a negative histological examination of the sBCC lesion at Week 10 (4 weeks post-treatment).
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 3% Active Cream BID: 3.0% active cream twice daily (BID)
- 3% Active Cream QD: 3.0% active cream once daily (QD) plus placebo cream QD
- Placebo BID: Placebo cream twice daily (BID)
Arm/Group | 3% Active Cream BID | 3% Active Cream QD | 1.5% QD | Placebo BID
Number analyzed (Participants) | 44 | 45 | 47 | 45
Participants | 9 | 5 | 7 | 9

2. Secondary Outcome: Number of Participants With Partial Response
Description: To determine the number of participants with a partial response, defined as a clinically significant decrease (ie, at least 50%) in the area of the sBCC lesion, computed as the product of the two principal diameters at Week 10 (4 weeks post-treatment)
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 3% Active Cream BID | 3% QD | 1.5% QD | Placebo BID
Number analyzed (Participants) | 46 | 45 | 48 | 45
Participants | 11 | 8 | 13 | 13

ADVERSE EVENTS:
Groups:
- 3% QD: 3.0% active cream once daily QD plus placebo cream QD
Arm/Group | 3% Active Cream BID | 3% QD | 1.5% QD | Placebo BID
Serious Adverse Events (participants affected / at risk) | 3/47 | 0/45 | 0/48 | 0/46
Other Adverse Events (participants affected / at risk) | 14/47 | 22/45 | 18/48 | 26/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3% Active Cream BID (N=47) | 3% QD (N=45) | 1.5% QD (N=48) | Placebo BID (N=46)
Blockage ( L ) Anterior Artery/Percutaneous Coronary Intervention (Stent) # 6 = Primary Care (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden Death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3% Active Cream BID (N=47) | 3% QD (N=45) | 1.5% QD (N=48) | Placebo BID (N=46)
Application Site Etythema (Skin and subcutaneous tissue disorders) | 8 (8) | 10 (10) | 8 (8) | 7 (7) — The most frequently reported treatment-emergent AE was application site erythema, which was reported in 33 of 186 subjects (17.7 %) in the overall safety population
Application Site Dryness (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Application Site Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Application site pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Application site bleeding (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes